CLINICAL TRIAL: NCT05271916
Title: An Open Label, Multicenter, Phase I/IIB Study of Dacomitinib Plus Anlotinib for Advanced Non-Small Cell Lung Cancer (NSCLC) Harboring Epidermal Growth Factor Receptor (EGFR) 21-L858R Mutations.
Brief Title: First-line Treatment With Dacomitinib Plus Anlotinib for Patients With Advanced NSCLC With EGFR 21L858R Mutations
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Baohui Han, Director of Respiratory Department, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IS22001
Record Dates: First submitted 2022-02-28; First posted 2022-03-09 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Non-Small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — dacomitinib

STUDY DESIGN:
Intervention Model Description: This is a multi-center, open-label, Phase I/IIB clinical study of Dacomitinib+Anlotinib in Advanced Non-Small Cell Lung Cancer (NSCLC) patients with EGFR 21L858R mutation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Combined treatment group (Experimental): Dacomitinib+Anlotinib: Patients will be treated with combined Dacomitinib and Anlotinib.
  Interventions: Drug: Dacomitinib+Anlotinib
- Dacomitinib monotherapy group (Active Comparator): Dacomitinib: Patients will be treated with Dacomitinib.
  Interventions: Drug: Dacomitinib

INTERVENTIONS:
Drug: Dacomitinib+Anlotinib — The dose of each drug in the combination Decomitinib and Anlotinib will be escalated or de-escalated until the recommended phase II dose (RP2D) is reached. Patients will then be treated with RP2D orally once a day.
  Arms: Combined treatment group
Drug: Dacomitinib — Dacomitinib orally on a continuous daily basis at a starting dose of 45 mg once a day until progressive disease.
  Arms: Dacomitinib monotherapy group

SUMMARY:
This is a multicenter, open label, Phase I/IIB study investigating the efficacy and safety of treatment with dacomitinib plus anlotinib as first-line therapy for patients with advanced non-small cell lung cancer (NSCLC) with epidermal growth factor receptor (EGFR) 21-L858R mutations. This study comprises two parts: 1. A dose escalation Phase I study to determine the recommended phase II dose. 2. a multi-center, open label, randomized controlled, Phase IIB study.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age and ≤75 years;
2. Provision of a voluntarily given, personally signed and dated, written informed consent document;
3. Histologically documented, unresectable, inoperable, locally advanced, recurrent or metastatic stage IIIB or IV non-small cell lung cancer (NSCLC);
4. It is acceptable for subjects with the presence of EGFR activating mutation (exon 19 deletion and the L858R mutation in exon 21) to be included in this Phase I study; Only subjects with the L858R mutation in exon 21 to be included in this Phase IIb;
5. At least one measurable disease by RECIST criteria version 1.1;
6. Patients with controlled or stable brain metastases;
7. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1, and life expectancy of at least 3 months;
8. No prior treatment with systemic therapy for advanced NSCLC, including TCM treatments;
9. Able to comply with required protocol procedures and able to receive oral medications;
10. Adequate organ function, including:

(1) Adequate bone marrow function Hemoglobin≥90g/L, absolute neutrophil count (ANC) should be ≥ 1.5x109/L, platelets should be ≥ 80x109/L; (2) Adequate liver function Total bilirubin ≤ 1.5 x upper normal limit (ULN), Aspartate Aminotransferase (AST) (SGOT) ≤ 2.5 x ULN (≤ 5.0 x ULN if hepatic metastases), Alanine Aminotransferase (ALT) (SGPT) ≤ 2.5 x ULN (≤ 5.0 x ULN if hepatic metastases), Creatinine≤ 1.5 x upper normal limit (ULN), or ≥ 60 mL/min; (3) Cardiac function: LVEF≥50% assessed by Doppler ultrasound；

Exclusion Criteria:

1. Small cell lung cancer (including mixed small cell and non-small cell lung cancer) and squamous cell carcinoma with cavitation;
2. Patients with concurrent EGFR T790M mutation or unknown mutation status or other mutation types;
3. Diagnosis of any other malignancy during the last 5 years, or with other malignancies at present;
4. Patients with pre-existing meningeal metastases;
5. Patients who have concurrent other malignant tumors;
6. Any history of hemoptysis, hematochezia, bloody sputum;
7. Tumor invasion or adjacent major vessels;
8. Patients with uncontrolled or significant systematic disease, including: active infection, thyroid dysfunction, uncontrolled hypertension, unstable angina pectoris, congestive heart failure, or myocardial infarction within 6 months, or severe arrhythmia requiring medication;
9. A history of other diseases, or metabolic dysfunction, or physical examination or laboratory results suggestive of a disease or condition that precludes the use of an investigational drug, or may affect the interpretation of the study results, or expose the patient to a high risk of treatment complications;
10. Any astrointestinal disorders resulting in inability to take medications orally, or requiring intravenous (IV) nutrition, or previous surgery impair drug absorption;
11. Pregnant or lactating females;
12. Patients allergic to any pharmaceutical ingredient.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-10-13 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Overall safety profile | Day 21 of Cycle 1, every 6 weeks until disease progression or death due to any cause, whichever occurred first (up to 22 months)
  Overall safety profile of combined Dacomitinib plus Anlotinib in Escalation Phase, including adverse events (AE), as defined and graded by the National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE 4.03], and first cycle Dose Limiting Toxicities (DLTs).
Progression Free Survival (PFS) | Day 21 of Cycle 1, every 6 weeks until disease progression or death due to any cause, whichever occurred first (up to 22 months)
  Progression Free Survival (PFS) is defined as the time from start of treatment to the date of disease progression as defined by RECIST v1.1 per investigator review or death due to any cause, whichever occurred first.

SECONDARY OUTCOMES:
Overall Survival (OS) | 48 months
  Overall Survival is defined as the time from start of treatment to the date of death for any cause. In the absence of confirmation of death, survival time will be censored at the last date the subject is known to be alive.
Best Overall Response (BOR) | From baseline until disease progression, up to 48 months
  Best overall response is best response from start of treatment until disease progression, and will calculated as the percentage of participants with an objective response (CR or PR) or stable disease, based on the RECIST v1.1, relative to the total number of participants enrolled in the cohort.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Wu YL, Cheng Y, Zhou X, Lee KH, Nakagawa K, Niho S, Tsuji F, Linke R, Rosell R, Corral J, Migliorino MR, Pluzanski A, Sbar EI, Wang T, White JL, Nadanaciva S, Sandin R, Mok TS. Dacomitinib versus gefitinib as first-line treatment for patients with EGFR-mutation-positive non-small-cell lung cancer (ARCHER 1050): a randomised, open-label, phase 3 trial. Lancet Oncol. 2017 Nov;18(11):1454-1466. doi: 10.1016/S1470-2045(17)30608-3. Epub 2017 Sep 25. PMID 28958502
- [Background] Mok TS, Cheng Y, Zhou X, Lee KH, Nakagawa K, Niho S, Lee M, Linke R, Rosell R, Corral J, Migliorino MR, Pluzanski A, Sbar EI, Wang T, White JL, Wu YL. Improvement in Overall Survival in a Randomized Study That Compared Dacomitinib With Gefitinib in Patients With Advanced Non-Small-Cell Lung Cancer and EGFR-Activating Mutations. J Clin Oncol. 2018 Aug 1;36(22):2244-2250. doi: 10.1200/JCO.2018.78.7994. Epub 2018 Jun 4. PMID 29864379
- [Background] Cheng Y, Mok TS, Zhou X, Lu S, Zhou Q, Zhou J, Du Y, Yu P, Liu X, Hu C, Lu Y, Zhang Y, Lee KH, Nakagawa K, Linke R, Wong CH, Tang Y, Zhu F, Wilner KD, Wu YL. Safety and efficacy of first-line dacomitinib in Asian patients with EGFR mutation-positive non-small cell lung cancer: Results from a randomized, open-label, phase 3 trial (ARCHER 1050). Lung Cancer. 2021 Apr;154:176-185. doi: 10.1016/j.lungcan.2021.02.025. Epub 2021 Feb 23. PMID 33721611
- [Background] Tabernero J. The role of VEGF and EGFR inhibition: implications for combining anti-VEGF and anti-EGFR agents. Mol Cancer Res. 2007 Mar;5(3):203-20. doi: 10.1158/1541-7786.MCR-06-0404. PMID 17374728
- [Background] Perdrizet K, Leighl NB. The Role of Angiogenesis Inhibitors in the Era of Immune Checkpoint Inhibitors and Targeted Therapy in Metastatic Non-Small Cell Lung Cancer. Curr Treat Options Oncol. 2019 Feb 18;20(3):21. doi: 10.1007/s11864-019-0617-6. PMID 30778772
- [Background] De Luca A, Carotenuto A, Rachiglio A, Gallo M, Maiello MR, Aldinucci D, Pinto A, Normanno N. The role of the EGFR signaling in tumor microenvironment. J Cell Physiol. 2008 Mar;214(3):559-67. doi: 10.1002/jcp.21260. PMID 17894407
- [Background] Saito H, Fukuhara T, Furuya N, Watanabe K, Sugawara S, Iwasawa S, Tsunezuka Y, Yamaguchi O, Okada M, Yoshimori K, Nakachi I, Gemma A, Azuma K, Kurimoto F, Tsubata Y, Fujita Y, Nagashima H, Asai G, Watanabe S, Miyazaki M, Hagiwara K, Nukiwa T, Morita S, Kobayashi K, Maemondo M. Erlotinib plus bevacizumab versus erlotinib alone in patients with EGFR-positive advanced non-squamous non-small-cell lung cancer (NEJ026): interim analysis of an open-label, randomised, multicentre, phase 3 trial. Lancet Oncol. 2019 May;20(5):625-635. doi: 10.1016/S1470-2045(19)30035-X. Epub 2019 Apr 8. PMID 30975627
- [Background] Zhou Q, Xu CR, Cheng Y, Liu YP, Chen GY, Cui JW, Yang N, Song Y, Li XL, Lu S, Zhou JY, Ma ZY, Yu SY, Huang C, Shu YQ, Wang Z, Yang JJ, Tu HY, Zhong WZ, Wu YL. Bevacizumab plus erlotinib in Chinese patients with untreated, EGFR-mutated, advanced NSCLC (ARTEMIS-CTONG1509): A multicenter phase 3 study. Cancer Cell. 2021 Sep 13;39(9):1279-1291.e3. doi: 10.1016/j.ccell.2021.07.005. Epub 2021 Aug 12. PMID 34388377
- [Background] Lin B, Song X, Yang D, Bai D, Yao Y, Lu N. Anlotinib inhibits angiogenesis via suppressing the activation of VEGFR2, PDGFRbeta and FGFR1. Gene. 2018 May 15;654:77-86. doi: 10.1016/j.gene.2018.02.026. Epub 2018 Feb 14. PMID 29454091
- [Background] Shen G, Zheng F, Ren D, Du F, Dong Q, Wang Z, Zhao F, Ahmad R, Zhao J. Anlotinib: a novel multi-targeting tyrosine kinase inhibitor in clinical development. J Hematol Oncol. 2018 Sep 19;11(1):120. doi: 10.1186/s13045-018-0664-7. PMID 30231931
- [Background] Han B, Li K, Wang Q, Zhang L, Shi J, Wang Z, Cheng Y, He J, Shi Y, Zhao Y, Yu H, Zhao Y, Chen W, Luo Y, Wu L, Wang X, Pirker R, Nan K, Jin F, Dong J, Li B, Sun Y. Effect of Anlotinib as a Third-Line or Further Treatment on Overall Survival of Patients With Advanced Non-Small Cell Lung Cancer: The ALTER 0303 Phase 3 Randomized Clinical Trial. JAMA Oncol. 2018 Nov 1;4(11):1569-1575. doi: 10.1001/jamaoncol.2018.3039. PMID 30098152
- [Background] Corral J, Mok TS, Nakagawa K, Rosell R, Lee KH, Migliorino MR, Pluzanski A, Linke R, Devgan G, Tan W, Quinn S, Wang T, Wu YL. Effects of dose modifications on the safety and efficacy of dacomitinib for EGFR mutation-positive non-small-cell lung cancer. Future Oncol. 2019 Aug;15(24):2795-2805. doi: 10.2217/fon-2019-0299. Epub 2019 Jul 17. PMID 31313942